CLINICAL TRIAL: NCT03758274
Title: Cognitive Behavioral Treatment by Phone to Promote Use of Alcohol Related Care and Reduce Drinking
Brief Title: Talk Therapy by Phone to Promote Treatment for Alcohol Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Medical University of South Carolina (Other); Syracuse University (Other)
Responsible Party: Principal Investigator, Kenneth Conner, Professor, Emergency Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSRB00072850; R01AA026815-01 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The University of Rochester based study team, led by MPI Conner, were masked to treatment assignment (which was performed at the Medical University of South Carolina), and the University of Rochester based team performed all follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Phone Intervention (Experimental): Cognitive-Behavioral Therapy for Treatment Seeking, CBT-TS, a manualized behavioral intervention, administered by telephone in a single session.
  Interventions: Behavioral: CBT by Phone to Promote Treatment
- Being Read A Pamphlet on Alcohol Treatment (Active Comparator): Guided review of a National Institute on Alcohol Abuse and Alcoholism (NIAAA) pamphlet on AUD treatment, administered by telephone in a single session.
  Interventions: Other: Reading the Subject a Pamphlet on Obtaining Alcohol Use Disorder Treatment

INTERVENTIONS:
Behavioral: CBT by Phone to Promote Treatment — Structured phone intervention to identify concerns about getting alcohol use disorder treatment and to work through those concerns using cognitive behavioral principles.
  Arms: CBT Phone Intervention
Other: Reading the Subject a Pamphlet on Obtaining Alcohol Use Disorder Treatment — The pamphlet was created by the National Institute on Alcohol Abuse and Alcoholism to describe evidence based treatments available for alcohol use disorder and how to obtain such treatment.
  Arms: Being Read A Pamphlet on Alcohol Treatment

SUMMARY:
A small percentage of individuals with alcohol use disorder (AUD) obtain alcohol-related care despite research showing that treatment is effective. This randomized controlled trial tests the efficacy of a brief, phone based cognitive behavioral intervention to increase treatment engagement, improve alcohol related outcomes, and show that treatment engagement is a mechanism for the improved outcomes in individuals with AUD.

ELIGIBILITY:
Inclusion Criteria:

* age 18-plus;
* score ≥ 16 on AUDIT;
* within the past 30 days, exceeding the limits for low-risk drinking adopted by NIAAA: >3 standard drinks on any occasion or >7 drinks per week (women); >4 drinks on any occasion or >14 drinks per week (men).

Exclusion Criteria:

* unable to communicate with the researcher in English;
* unable to comprehend the nature of the study;
* history of alcohol-related care;
* alcohol withdrawal necessitating medical evaluation;
* residency outside of The Greater Rochester Area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT Phone Intervention | Being Read A Pamphlet on Alcohol Treatment
Started | 197 | 203
Completed | 186 (3-month follow-up) | 190 (3-month follow-up)
Not Completed | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT Phone Intervention | Being Read A Pamphlet on Alcohol Treatment | Total
Number analyzed (Participants) | 197 | 203 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.5) | 41.1 (10.9) | 40.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 92 | 199
  Male | 90 | 111 | 201
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 158 | 159 | 317
  Black | 26 | 27 | 53
  Asian | 3 | 6 | 9
  Native American-Alaskan Native | 1 | 1 | 2
  More than one race | 8 | 8 | 16
  Other race | 1 | 2 | 3
  Hispanic ethnicity (across races) | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 197 | 203 | 400
Average Drinks Per Drinking Day (in past 30 days) [Mean (Standard Deviation); unit: standard drinks] | 6.7 (3.7) | 6.7 (3.5) | 6.7 (3.6)
Days Abstinent (in past 30 days) [Mean (Standard Deviation); unit: days (scale 0-30)] | 8.5 (7.7) | 8.1 (7.3) | 8.3 (7.5)
Number Initiating Alcohol Use Disorder Treatment [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Drinks Per Drinking Day
Description: Average number of standard drinks on days of alcohol consumption at 3-month follow-up
Time Frame: prior 30 days (at 3-month follow-up)
Measure: Mean (Standard Deviation); unit: drinks per occasion
Arm/Group | CBT Phone Intervention | Being Read A Pamphlet on Alcohol Treatment
Number analyzed (Participants) | 197 | 203
drinks per occasion | 5.5 (3.8) | 5.4 (3.5)
Statistical Analysis 1: Comparison: CBT Phone Intervention vs Being Read A Pamphlet on Alcohol Treatment; Test type: Superiority; p = 0.746, Based on simple path model in Mplus

2. Primary Outcome: Days Abstinent
Description: Number of days abstinent from alcohol use in prior 30 days
Time Frame: prior 30 days (at 3-month follow-up)
Measure: Mean (Standard Deviation); unit: Days abstinent (in past 30 days)
Arm/Group | CBT Phone Intervention | Being Read A Pamphlet on Alcohol Treatment
Number analyzed (Participants) | 197 | 203
Days abstinent (in past 30 days) | 15.5 (10.5) | 14.6 (9.9)
Statistical Analysis 1: Comparison: CBT Phone Intervention vs Being Read A Pamphlet on Alcohol Treatment; Test type: Superiority; p = 0.247, Based on simple path model in Mplus

3. Primary Outcome: Number Initiating Alcohol Use Disorder Treatment
Description: Number Attending any Alcohol Use Disorder Treatment Session(s) over 3-month follow-up
Time Frame: over 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CBT Phone Intervention | Being Read A Pamphlet on Alcohol Treatment
Number analyzed (Participants) | 197 | 203
Participants | 38 | 36
Statistical Analysis 1: Comparison: CBT Phone Intervention vs Being Read A Pamphlet on Alcohol Treatment; Test type: Superiority; p = 0.689, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CBT Phone Intervention | Being Read A Pamphlet on Alcohol Treatment
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/203
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/203
Other Adverse Events (participants affected / at risk) | 0/197 | 1/203
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT Phone Intervention (N=197) | Being Read A Pamphlet on Alcohol Treatment (N=203)
Acute alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) — Acute alcohol withdrawal requiring alcohol detoxification

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03758274/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03758274/SAP_001.pdf